CLINICAL TRIAL: NCT06187935
Title: Early Adjuvant Diagnosis Clinical Trial of Pulmonary Nodules Based on Circulating Tumor Cells.
Brief Title: Early Adjuvant Diagnosis of Pulmonary Nodules Based on CTC.
Status: Completed | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Guangying Zhu, chief physician, China-Japan Friendship Hospital
Other Study IDs: 2018-170-K124
Record Dates: First submitted 2023-12-07; First posted 2024-01-03 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Nodules, Solitary; Pulmonary Nodules, Multiple
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — circulating tumor cell
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- pulmonary nodule group: Patients with pulmonary nodules no more than 3cm on CT imaging.

SUMMARY:
The goal of this observational clinical trial is to evaluate the value of circulating tumor cell detection in the early diagnosis of malignant pulmonary nodule. The main questions it aims to answer is: the sensitivity and specificity of peripheral blood circulating tumor cell detection in differentiating benign and malignant pulmonary nodules (≤3cm). Participants will be asked provide 4mL of peripheral blood for the test.

DETAILED DESCRIPTION:
The aim of this clinical trial is to evaluate the value of circulating tumor cell detection in the early diagnosis of malignant pulmonary nodule. Patients with clinical suspected malignant pulmonary nodules will be included in this trial. Peripheral blood of participants will be collected before surgery or biopsy. Clinical and imaging data of enrolled patients will also be collected. Pathological diagnosis is the gold standard for differentiating benign and malignant pulmonary nodules. The sensitivity and specificity of CTC detection for diagnosing malignant pulmonary nodules will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with single or multiple pulmonary nodules on CT imaging; 2. Subjects ≥18 years old, regardless of gender, occupation, and region, should have independent capacity for civil conduct and sign the informed consent for clinical study; 3. Subjects are generally in good condition, with ECOG score 0-1 and life expectancy of no less than 2 months; 4. Organ function level requirements:

1. Peripheral blood: 1.5 x 10^9/L≤ absolute neutrophil count (ANC) ≤15 x 10^9/L, platelets ≥100 x 10^9/L, hemoglobin ≥9.0 g/dL; Prothrombin time (PT) ≥11 seconds, International normalized ratio (INR) ≥0.8;
2. Bilirubin ≤1.5 times the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times the upper limit of normal;
3. Serum creatinine ≤1.5 times the upper limit of normal value.

Exclusion Criteria:

1. The subjects had a history of malignant tumors, or serious cardiovascular and cerebrovascular diseases (had undergone heart stent surgery within 6 months or had been admitted to ICU, CCU or other intensive care units due to cardiovascular and cerebrovascular diseases, or EF≤50%); b. Severe vasculopathy, pulmonary tuberculosis or large-scale acute inflammation (including but not limited to acute bronchitis, vasculitis, etc.) or active chronic infection (HIV, HBV, HCV, etc.) within 3 months; 3. Poor compliance, unable to cooperate with the research program; 4. Participants in any drug trial within three months prior to enrollment; 5. Pregnant or breastfeeding; 6. Puncture/Surgical contraindications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary nodules no more than 3cm on CT imaging that are clinically suspected to be malignant and scheduled for surgery or biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
sensitivity | until the samples are collected and tested as planned, up to 72 months
  the ability of peripheral blood CTC count detection to identify malignant pulmonary nodules when the real condition is malignancy
specificity | until the samples are collected and tested as planned, up to 72 months
  the ability of peripheral blood CTC count detection to exclude malignant pulmonary nodules when the real condition is benign disease

CONTACTS AND LOCATIONS:
Overall Officials: Guangying Zhu, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Original research data including study protocol and statistical analysis plan will be shared after the study is completed and the research results are published.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available starting 6 months and ending 5 years following article publication.
Access Criteria: People who provide reasonable research protocols can get access to the data by contacting the researchers.